CLINICAL TRIAL: NCT03015922
Title: VIRel: Viral Immunotherapy in Relapsed/Refractory Multiple Myeloma - A Phase I Study to Assess the Safety and Tolerability of REOLYSIN® (Pelareorep) in Combination With Lenalidomide or Pomalidomide
Brief Title: Viral Immunotherapy in Relapsed/Refractory Multiple Myeloma
Acronym: MUKeleven
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Leeds (Other)
Collaborators: Myeloma UK (Other); Oncolytics Biotech (Industry); Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Gordon Cook, Consultant Haematologist, The Leeds Teaching Hospitals NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM16/118
Record Dates: First submitted 2016-11-16; First posted 2017-01-10 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; pomalidomide; reolysin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenalidomide or pomalidomide, plus REOLYSIN (Experimental): Lenalidomide capsules, oral, maximum 10mg daily on days 1-21 of 28-day cycles. OR Pomalidomide capsules, oral, maximum 1mg daily on days 1-21 of 28-day cycles.
  Plus (all patients):
  REOLYSIN® , intravenous infusion, maximum 3x10^10 TCID50 on days 1, 8, 15 and 22 of 28-day cycles.
  Interventions: Drug: Lenalidomide or Pomalidomide; Biological: REOLYSIN

INTERVENTIONS:
Drug: Lenalidomide or Pomalidomide — Patients will received either lenalidomide or pomalidomide, depending on which drug they were receiving prior to the trial (they will receive the same as before).
Biological: REOLYSIN — Patients will receive Reolysin alongside either lenalidomide or pomalidomide
  Other Names: Pelareorep; Reovirus

SUMMARY:
This study will recruit patients currently receiving either lenalidomide or pomalidomide whose disease is relapsing. This is a dose escalation study and the aim is to determine the maximum tolerated dose (MTD) of REOLYSIN® that can be given in combination with lenalidomide or pomalidomide. The study will also investigate the safety, side effects and effectiveness of this treatment combination. Pomalidomide and lenalidomide will be evaluated separately as two separate groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with symptomatic multiple myeloma (according to IMWG 2014 criteria)
* Evaluable disease by modified IMWG criteria (i.e. by abnormal serum M protein, urinary M protein or serum free light chain assays)
* Currently receiving either lenalidomide or pomalidomide therapy, alone or in combination with other myeloma therapy, with evidence of serological or clinical disease progression as defined by IMWG criteria (2011)
* Life expectancy of ≥ 3 months
* ECOG performance status of ≤2
* Required laboratory values within 14 days prior to dose allocation:
* Absolute neutrophil count ≥ 1.0 x10^9 /L. (growth factor support is not permitted)
* Platelet count ≥ 70 x 10^9/L. (platelet support is not permitted; platelets < 70 but ≥ 25 acceptable if bone marrow is > 50% infiltrated by MM)
* Haemoglobin ≥ 8 g/dL. Blood support is permitted
* Serum bilirubin ≤ 2 x upper limit of normal (ULN)
* ALT or AST ≤ 2.5 x ULN
* Serum creatinine ≤ 2 x ULN
* Corrected calcium ≤ 2.8 mmol/l
* Negative HIV and viral (B and C) hepatitis test result within 14 days prior to dose allocation
* Able to give informed consent and willing to follow trial protocol
* Aged 18 years or over
* All participants must agree to follow the Celgene Pregnancy Prevention Programme (PPP) and participate in the counselling associated with this:
* Females of childbearing potential (FCBP) must agree to utilise two reliable forms of contraception simultaneously or practice complete abstinence for at least for 28 days prior to starting trial treatment, during the trial and for at least 28 days after trial treatment discontinuation, and even in case of dose interruption, and must agree to Celgene PPP pregnancy testing during this timeframe
* Females must agree to abstain from breastfeeding during trial participation and 28 days after trial drug discontinuation
* Males must agree to use a latex condom during any sexual contact with FCBP (or must practice complete abstinence) during the trial, including during dose interruptions and for 28 days following discontinuation from this trial even if he has undergone a successful vasectomy
* Males must also agree to refrain from donating semen or sperm while on pomalidomide including during any dose interruptions and for 28 days after discontinuation from this trial
* All participants must agree to refrain from donating blood while on trial drug including during dose interruptions and for 28 days after discontinuation from this trial

Exclusion Criteria:

* Non-secretory multiple myeloma
* Pregnant (positive pregnancy test) in line with the Celgene Pregnancy Prevention Programme or breast feeding
* Previous anti-tumour therapies including experimental agents, other than lenalidomide or pomalidomide, within 28 days of the start of protocol treatment. Steroid therapy is permitted, but must be stopped 48 hours prior to cycle 1 day 1
* Concurrent or previous malignancies (<12 months post end of treatment) at other sites, with the exception of appropriately treated localised epithelial skin or cervical cancer, or incidental histologic findings of prostate cancer (TNM stage T1a or 1b). Participants with histories (≥12 months) of other tumours, in remission and not currently on therapy, may be entered
* System corticosteroid therapy for comorbidities (i.e. medical conditions other than multiple myeloma) that cannot be stopped for the duration of the trial. Topical corticosteroid therapy is not an exclusion criterion.
* Any history of known hypersensitivity to any of the trial medications or excipients
* Active symptomatic fungal, bacterial, and/or viral infection
* Poorly controlled or serious medical or psychiatric illness that, in the Investigator's opinion, is likely to interfere with participation and/or compliance in this clinical trial
* Patients with significant cardiovascular disease (e.g. history of congestive heart failure requiring therapy (≥ NYHA Class III), presence of severe valvular heart disease, presence of an atrial or ventricular arrhythmia requiring treatment, uncontrolled hypertension, or history of QTc abnormalities)
* Radiotherapy or major surgery within 4 weeks prior to registration
* Greater than or equal to grade 2 neuropathy, with or without pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities | After cycle 1 (28 days) of treatment. Assessed in real-time for each patient to inform dose escalation decisions.
  Dose-limiting toxicities (DLTs), within the first cycle (until cycle 2, day 1), in order to establish the Maximum Tolerated Dose (MTD) of REOLYSIN® in combination with lenalidomide or pomalidomide, in two separate groups of participants.

SECONDARY OUTCOMES:
Safety profile of REOLYSIN® and lenalidomide | Until 28 days after the last dose of trial treatment for each patient. Assessed up to 27 months.
  Safety will be reported based on the occurrence of SAEs, SARs and SUSARs.
Safety profile of REOLYSIN® and pomalidomide | Until 28 days after the last dose of trial treatment for each patient. Assessed up to 27 months.
  Safety will be reported based on the occurrence of SAEs, SARs and SUSARs.
Toxicity profile of REOLYSIN® and lenalidomide | Until 28 days after the last dose of trial treatment fior each patient. Assessed up to 27 months.
  Toxicity will be reported based on adverse events, as graded by CTCAE V4.0, and determined by routine clinical assessments at each centre.
Toxicity profile of REOLYSIN® and pomalidomide | Until 28 days after the last dose of trial treatment fior each patient. Assessed up to 27 months.
  Toxicity will be reported based on adverse events, as graded by CTCAE V4.0, and determined by routine clinical assessments at each centre.
Response rate (stable disease or better) after 6 cycles of therapy | Data will be collected from each patient after they have received 6 cycles of therapy, if this stage is reached. 6 cycles are expected to take 24 weeks to complete.
  Measured only in patients treated at the maximum tolerated dose
Maximum response within 6 cycles of therapy | Assessed for each patient after they have received 6 cycles of treatment. 6 cycles are expected to take 24 weeks to complete.
  Measured only in patients treated at the maximum tolerated dose
Maximum response overall | Assessed for each patient after they have completed treatment on the trial. Assessed up to 27 months.
  Measured only in patients treated at the maximum tolerated dose
Time to maximum response | Assessed for each patient after they have completed treatment on the trial. Assessed up to 27 months.
  Measured only in patients treated at the maximum tolerated dose
Progression-free survival | Calculated for each patient from the date of registration up to first documented evidence of disease progression or death. Assessed up to 27 months.
  Measured only in patients treated at the maximum tolerated dose. Participants who have not progressed at the time of analysis will be censored at the last date they were known to be alive and progression free.
Overall survival | Calculated for each patient from the date of registration to death. Assessed up to 27 months.
  Measured only in patients treated at the maximum tolerated dose. Participants who have not died at the time of analysis will be censored at the last date they were known to be alive.

OTHER OUTCOMES:
Immune response biomarker profile of REOLYSIN and lenalidomide administered in combination | This will be assessed based on samples taken throughout each patient's time on the trial. Assessed up to 27 months.
  Biomarker profiling of the combination treatment
Immune response biomarker profile of REOLYSIN® and pomalidomide administered in combination | This will be assessed based on samples taken throughout each patient's time on the trial. Assessed up to 27 months.
  Biomarker profiling of the combination treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Cook, Principal Investigator — St. James's University Hospital
Locations (2):
- United Kingdom (2):
  - St James's University Hospital, Leeds
  - Sheffield Teaching Hospitals NHS Foundation Trust, Northern General Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No